CLINICAL TRIAL: NCT06674668
Title: Immediate Effect of Wearable Vibrotactile Stimulation on Pain and Sense in Patients with Lateral Epicondylitis
Brief Title: Effect of Vibrotactile Stimulation in Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Istanbul Kültür University (Other)
Responsible Party: Principal Investigator, Imge NAS, Lecturer, Istanbul Kültür University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: İK-2023-01
Record Dates: First submitted 2024-10-21; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Lateral Epicondylitis; Vibration Therapy; Physiotherapy
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention includes traditional physiotherapy and vibrotactile device use.
  Interventions: Other: Vibrotactile stimulation
- Control group (Active Comparator): For traditional physiotherapy, passive stretching exercises, radial head mobilization and deep friction massage will be applied to the affected extremity.
  Interventions: Other: Traditional physiotherapy

INTERVENTIONS:
Other: Vibrotactile stimulation — The intervention includes traditional physiotherapy and 20 minutes of vibrotactile device use. As traditional physiotherapy, 30 seconds of 8 repetitions of passive wrist stretching exercises, radial head mobilization and deep friction massage will be applied to the affected extremity. Afterwards, the Intellinetix Elbow Wearable Vibration Device providing vibration will be worn on the affected tissue. The patient will remain in a comfortable position on the treatment table with the affected extremity for 20 minutes (10 minutes × 2).
  Arms: Intervention group
Other: Traditional physiotherapy — For traditional physiotherapy, passive stretching exercises, radial head mobilization and deep friction massage will be applied to the affected extremity. Stretching exercises will be performed on the wrist flexor and extensor muscles for 30 seconds and 8 repetitions. Mill's manipulation, described by James Cyriax, will be applied once for radial head mobilization. The treatment will be completed with a 5-minute deep friction massage, affecting the wrist extensor muscle tendons and their ending points.
  Arms: Control group

SUMMARY:
It is aimed to investigate the immediate effect of vibrotactile stimulation on pain, sense and functionality in patients with lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) is a chronic degenerative disease of the attachment site of the extensor tendons to the lateral epicondyle of the humerus. The annual incidence is 1-3% of the world population and is most common between the ages of 30 and 60. Although LE is often called "tennis elbow," a small percentage of patients play tennis. The etiology of the disease is multifactorial, and it is generally thought to be caused by repetitive wrist activities that include gripping, wrist extension, and supination. Most patients recover spontaneously within 1-2 years. However, loss of work capacity is quite common in jobs that require the use of the upper extremity.

The pathophysiology of the disease is currently explained by degenerative mechanisms instead of the idea of inflammatory infiltration. Microtears and tendinosis caused by increased force on the tendon are supported by ultrasonographic examinations. However, currently, pain and functional disability in daily life are explained by sensory changes such as pain pressure threshold, impaired vibration perception and joint position sense rather than tendon structure changes. Clinically, lateral elbow pain results in decreased grip strength and proprioception, and consequently loss of function.

In LE management, the aim is to relieve pain, minimize excessive loads on the arm and restore the patient to optimal daily life activities and former functionality.

While there is insufficient evidence on the effectiveness of surgical interventions in treatment, nonoperative methods are frequently preferred. Patient education, use of splints, medical treatments, biological treatments, physical agents, taping, and manual therapy approaches are frequently used. While conservative treatments remain up-to-date for pain and disability, the most appropriate treatment strategy is controversial.

The use of technology in physiotherapy has been increasing in recent years. In addition to motor movement, the development of sensory skills is also emphasized. On the other hand, vibrotactile stimulation has been reported to contribute to the sensory processing mechanism by causing different activity levels in the brain. There are no studies in the literature investigating the effects of wearable vibration technology on sensory parameters in LE patients. The aim of this study is to investigate the effects of wearable vibrotactile application on pain, sensation and upper extremity function compared to traditional physiotherapy in patients with LE.

Patients diagnosed with LE will be included in the study. Participants will be randomized into two groups. Patients in both groups will receive one session of conventional physiotherapy on the affected extremity. In addition to the intervention group, the use of a wearable vibrotactile device will be provided. Immediate effects will be evaluated before and after the application in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age
* Patients diagnosed with lateral epicondylitis

Exclusion Criteria:

* Having had elbow surgery
* Having a history of congenital or acquired orthopedic, neurological, or rheumatological conditions affecting the upper limb
* Having received any conservative treatment for the diagnosis of lateral epicondylitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | from pre-interventional time to post-interventional about 1st hour
  A 10 cm visual analog scale (VAS) was used to assess pain intensity. A horizontal 10 cm ruler was used (0 = no pain and 10 = worst pain).
Pressure pain threshold | from pre-interventional time to post-interventional about 1st hour
  The J tech brand algometer device will be used for the pressure pain threshold measurement. The trigger points will be found by palpation. The person will be told that the device will apply pressure to the trigger point and that they will give the command "stop" when they first feel the pain.
Joint position sense | from pre-interventional time to post-interventional about 1st hour
  Elbow joint position sense will be measured with an inclinometer for 45 and 60 degree flexion target angle. The elbow will be brought to the target angle and they will be asked to memorize the movement by holding it for 10 seconds. Then, they will be asked to bring the target force they learned themselves. The absolute value of the difference between the target value and the last measurements will be taken as the error score.

SECONDARY OUTCOMES:
Hand grip sensitivity level | from pre-interventional time to post-interventional about 1st hour
  Pneumatic dynamometer will be used for measurement. The individual's maximum grip strength will be measured and half will be taken to determine the target strength. First, the target strength measurement will be made, then the target measurement will be asked to repeat it without seeing the target measurement value. The absolute value of the difference between the targeted value and the measurements will be calculated and recorded as an error score.
Grip Strength | from pre-interventional time to post-interventional about 1st hour
  Takei Hand Grip Dynamometer will be used to assess painless grip strength. Subjects will be instructed to increase their grip strength and stop if they feel pain or discomfort. Painless grip strength will be measured 3 times with 30 seconds between measurements and an average score will be obtained.
Functional assessment | 2 weeks
  The Turkish version of the Disability Score for the Arm, Shoulder and Hand (DASH) will be used to assess upper extremity physical function. The questionnaire consists of 30 questions. Scores range from 0 to 100. Higher scores indicate lower functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kultur University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No